CLINICAL TRIAL: NCT01692405
Title: Semi-automatic Download of Prostate Biopsy Cores While Keeping the Orientation, Unfolding and Unity of the Sample
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UC Care, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 0086-12-EMC
Record Dates: First submitted 2012-09-12; First posted 2012-09-25 (Estimated); Last update posted 2019-04-19 (Actual); Status verified 2012-09

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard method (No Intervention): Standard method- shaking the biopsy needle into a formalin container.
- Download onto a biopsy sponge pad (Active Comparator): Samples will be downloaded by moving the needle notch on a biopsy sponge pad.
  Interventions: Procedure: biopsy sponge pad
- Dowloading the biopsy cores using NavigoBx system (Experimental): Downloading the biopsy cores using NavigoBx™ system. The NaviGoBx™ device is intended for the retention of a biopsy specimen and for preservation of the specimen's in-needle location and orientation.
  Interventions: Device: NaviGo Bx™

INTERVENTIONS:
Device: NaviGo Bx™ — The NaviGoBx™ system is a device and method that enables an accurate reporting of the exact longitudinal location and direction of the biopsy specimen along the needle notch as well as the accurate length of the specimen. Acquiring this information during the biopsy extraction session provides an accurate designation of the location of any later region of interest within the specimen itself to the longitudinal position along the needle mandrel.
  Arms: Dowloading the biopsy cores using NavigoBx system
Procedure: biopsy sponge pad — the biopsy core is downloaded onto a biopsy sponge pad which is than entered into a biopsy cassette.
  Arms: Download onto a biopsy sponge pad

SUMMARY:
Performance evaluation of a novel, semi-automated device and method for needle core biopsy download compared to standard methods in terms of:

1. Biopsy core length obtained (i.e. collecting all tissue fragments)
2. Biopsy core yield (i.e. percent of tissue loss during the pathologic processing)
3. Pathologist interpretability
4. Processing time
5. Prostate cancer detection.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Planned for radical or open prostatectomy operation or Planned for TRUS prostate biopsy procedure.
* Signed informed consent.

Exclusion Criteria:

* Patient's unwilling to participate.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 436 (Actual)
Dates: Start 2013-04-29 (Actual); Primary Completion 2017-04-05 (Actual); Study Completion 2017-04-24 (Actual)

PRIMARY OUTCOMES:
percent of tissue loss | 1 year
  percent of biopsy tissue loss during pathologic processing. comparing the core length as recorded on the biopsy needle notch and on the histology slide

SECONDARY OUTCOMES:
prostate cancer detection rate | 1 year
processing time | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Haemek madical center, Afula, Israel

REFERENCES:
- [Background] Obek C, Doganca T, Erdal S, Erdogan S, Durak H. Core length in prostate biopsy: size matters. J Urol. 2012 Jun;187(6):2051-5. doi: 10.1016/j.juro.2012.01.075. Epub 2012 Apr 11. PMID 22498214